CLINICAL TRIAL: NCT03234946
Title: Effect of the CAIPaDi Care Model in Relatives of Patients With Type 2 Diabetes Mellitus
Acronym: CAIPaDi
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Collaborators: Mexican National Institute of Public Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2145
Record Dates: First submitted 2017-07-27; First posted 2017-08-01 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Metabolic Syndrome
Keywords: Diabetes; Family; Impaired fasting-glucose; Carbohydrate intolerance
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus; Glucose-Galactose Malabsorption

STUDY DESIGN:
Intervention Model Description: Relatives of CAIPaDi patients that present on their initial evaluation either overweight, obesity, hypertension, glucose intolerance and/or secondary dyslipidemia will be invited to participate.
  Those who accept will require to attend the center twice. On the first visit, an anthropometric evaluation and laboratory studies will be performed; an oral glucose tolerance (OGTT) test will be carried out if the glucose value is over 100 mg/dl. If the OGTT results are abnormal, the individual will be included in the study sample.
  Those who have an abnormal OGTT and are included in the study sample will be randomized into two groups.
  The change of the main variables (weight, waist circumference, serum glucose, glycated hemoglobin, blood pressure, triglycerides and non-HDL cholesterol) will be assessed 3 months later, along with the effect on patients with diabetes parameters.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (No Intervention): Relatives of patients with diabetes who will only attend sessions at the center along with the patients on all the interventions of the center (except psychology and psychiatry), receiving instructions from each area on the first and fourth visit. When the patient with diabetes is in the psychology or psychiatry consultation, the relative will also be evaluated in these areas in an analogue form.
- Group B (Experimental): Relatives who will receive multidisciplinary care at the center The subjects from group B will be asked to be accompanied by another relative. If they accept, they will be included as a patient of the CAIPaDi program to receive all the interventions of the second, third and fourth visits in an individual form, without following the patient with diabetes.
  Interventions: Behavioral: CAIPaDi

INTERVENTIONS:
Behavioral: CAIPaDi — Patients are attended in 1 day by 9 specialists (endocrinologist, diabetes educators, nutritionist, psychologist, physical activity specialist, foot care and ophthalmologist). They are attended in 4 monthly visits. After the initial phase, patients come back to the Center at 1 and 2 years for evaluation and reinforcement
  Arms: Group B

SUMMARY:
Diabetes is a chronic disease that requires long-term lifestyle changes that may affect the whole family. Hence, during the last decade, studies have focused mainly in the role of the members of the family and their influence in life quality or clinical outcomes of patients with diabetes. Therefore, the delivery of education only to the patients with type 2 diabetes mellitus may restrict the expectations of success in achieving the necessary modifications in lifestyle.

Objectives: To assess the effect of the CAIPaDi (Centre of Comprehensive Care for the Patients with Diabetes) program interventions on various health indicators relatives of patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Diabetes mellitus is one of the most challenging health issues of our time, the percentage of adults with this disease tripled in Mexico between 1993 and 2012; In 1993 the prevalence was 6.7% (cases previously diagnosed 4.6% and diagnosed during the survey 2.1%), whereas in 2012, the prevalence was 14.4% (7.3% previously diagnosed and 7.1% diagnosed during the survey) Identifying individuals at risk for developing diabetes and implementing prevention strategies is the optimal solution. Carbohydrate intolerance and impaired fasting glucose raise the risk of developing diabetes up to 20 times compared to those with normal levels of HbA1C and a progression rate to diabetes of 10% per year in the absence of any intervention.

Randomized studies have shown that progression from impaired fasting glucose and glucose intolerance to type 2 diabetes mellitus and its complications can be prevented by interventions focused on changes in lifestyle. This contributed to the implementation of new guidelines for the management of prediabetes, emphasizing the importance of timely interventions in this condition, which may be the most cost-effective alternative to avoid complications.

One of the most important studies in primary diabetes prevention, the Diabetes Prevention Program (DPP), provided scientific evidence on the prevention and delay in the onset of diabetes in high-risk individuals, with a 58% risk reduction through lifestyle modifications, such as reduced fat and calorie intake, increased physical activity up to at least 150 minutes per week and loss of 5-7% of body weight.

Another multicenter, randomized trial, the Finnish Diabetes Prevention Study (DPS), showed that type 2 diabetes is preventable with lifestyle multidisciplinary interventions, with a 58% risk reduction similar to that of the DPP study in the group who received intensive treatment, compared to the control group, even significant changes were observed in metabolic parameters one and three years afterwards.

In addition, a randomized, multicenter study in the city of Da Qing, China, with a population of 110,660 participants, demonstrated that diet and / or exercise lead to a significant decrease in the incidence of diabetes over a 6-year period in patients with carbohydrate intolerance, with an incidence of 67.7% in the control group, 43.8% in the group undergoing dietary changes and 46% in the diet and exercise group.

Family history of diabetes is an independent risk factor for having the disease and provides information for the screening of individuals at risk and even represents an even more sensitive indicator than the presence of obesity.

Diabetes is a chronic disease that involves changes in the patient's lifestyle that can affect the whole family. During the last decade, studies have focused mainly on the role of family members and their influence on the quality of life or clinical course of patients with diabetes. Therefore, providing education only to the individual diagnosed with type 2 diabetes could restrict the chances of success in achieving the necessary changes in lifestyle.

Some studies have shown that the familial nature of type 2 diabetes is manifested by the presence of insulin resistance in first-degree relatives without diabetes, while others have revealed B-cell dysfunction, it seems that both insulin resistance and a diminished B-cell compensation are the family metabolic phenotype of type 2 diabetes mellitus. This highlights the importance of providing diabetes education not only to the patient, but also to their relatives, especially those who already have additional risk factors or prediabetes.

In cross-sectional studies of diabetes, social support has been associated with a better glycemic control in type 2 diabetes and is positively related to overall health status and lifestyle changes. Additionally, the health status of family members of patients attending the sessions has been demonstrated, and social and family support in general is positively linked to health status and transcendental changes in lifestyle.

These findings are justified by the results of the second multinational study, Diabetes Attitudes, Wishes and Needs (DAWN2TM), in which the disease was studied from the perspective of family members, patients and health professionals. Family members who deemed a greater responsibility for the management of diabetes had a lower quality of life and higher levels of disease impact and perceived burden, while less responsibility for the management of diabetes perceived by the patient's family members and an effective collaboration among them correlates with improved psychological well-being and quality of life for family members.

Diabetes is associated with a sense of social disadvantage and stress not only in patients with diabetes but also in the members of their family, so there is a need to foster a larger network of family support through educational programs and to involve them in the treatment of the illness.

To date there are no studies that accurately analyze the impact of social support on maintaining lifestyle changes in a supportive group setting.

The study Families United analyzed the effect of social support in the prevention of diabetes, which has proved to be important for its management and even for other diseases such as obesity, it has been used to convey information regarding prevention of diabetes to minority and high-risk groups in communities.

The social context in which the patient carries out self-care activities determines its success, so that obstructive behaviors such as sabotage or underestimating the patient's effort or hampering their self-care are associated with a greater HbA1C and a reduction of motivation and adherence to treatment, diet plan and exercise.

Despite the high prevalence of obstructive behaviors among relatives of patients with diabetes, few interventions focus on the negative aspects of family interactions.

Family support behaviors or sabotage in diabetes have been independently associated with adherence to self-care behavior and glycemic control among adults with diabetes and low sociocultural level. DAWN-II found that more than one-third of family members wish to be more involved in managing the patient's disease.

A study was conducted in 2013 based on socio-cognitive theory, which focuses on the influence of the social environment (family members) on changes in health habits to overcome barriers to self-management of diabetes and improve self-efficacy. With a population of 36 patients and 37 relatives, with a duration of 14.6 months. The intervention consisted of 2 family sessions and 8 weekly group educational sessions for participants and their families. It was possible to demonstrate positive effects on systolic blood pressure, knowledge of diabetes, self-efficacy, self-management of general and specific diet, glucose monitoring, foot care, fruit and vegetable consumption and physical and mental components associated with quality of life in the participants. There was also a significant improvement in BMI and knowledge of diabetes in family members, suggesting that a culturally-tailored diabetes education program provides a significant benefit to both Hispanic patients with diabetes and their families. In addition, it has been observed that total family involvement in diabetes education helps to increase knowledge, attitude and practice scores in patients with type 2 diabetes mellitus and to improve their quality of life, with significant effects on glycemic control and weight.

For this reason, a collaborative therapeutic partnership between the patient, his family and health care providers is essential, encouraging family members to participate in programs to avoid patient isolation, maintaining family cohesion and promoting health behaviors that reduce the risk and early onset of diabetes in family members.

ELIGIBILITY:
Inclusion Criteria:

* Being a relative of a patient of CAIPaDi
* Fasting glucose of <125 mg/dl
* Serum glucose of <199 mg/dl 2 hours after a glucose load of 75 gr

Exclusion Criteria:

* Diagnosis of diabetes
* Smoking
* Who has any disabling or priority health condition other than prevention of diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Estimated)
Dates: Start 2017-06-19 (Actual); Primary Completion 2021-06-19 (Estimated); Study Completion 2021-06-19 (Estimated)

PRIMARY OUTCOMES:
Glycated hemoglobin | 1 year
  60% of patients with a glycated hemoglobin of <5.8
Body Mass Index | 1 year
  Difference of 2kg/m2 between groups

SECONDARY OUTCOMES:
Serum glucose | 1 year
  <126 mg/dl
Non-HDL cholesterol | 1 year
  <160
Triglycerides | 1 year
  <150
Blood pressure | 1 year
  <140/90 mmHg
Weight loss | 1 year
  5% reduction of basal weight
Waist circumference | 1 year
  5 cm reduction of basal waist circumference
Hospital Anxiety and Depression Scale (HAD) | 1 year
  score of <7 points
Minutes of exercise per day | 1 year
  >30 minutes of exercise per day
Steps per day | 1 year
  >10,000 steps per day

CONTACTS AND LOCATIONS:
Overall Officials: Ana C García Ulloa, MD, Principal Investigator — Grade A Specialized Physician
Locations (2):
- Mexico (2):
  - Instituto Nacional de Salud Pública, Cuernavaca, Morelos
  - Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Villalpando S, Shamah-Levy T, Rojas R, Aguilar-Salinas CA. Trends for type 2 diabetes and other cardiovascular risk factors in Mexico from 1993-2006. Salud Publica Mex. 2010;52 Suppl 1:S72-9. doi: 10.1590/s0036-36342010000700011. PMID 20585732
- [Background] Aguilar Salinas CA, Gómez Diaz RA, Gomez Perez FJ. Type 2 diabetes in Mexico: Main Challenges and possible solutions. Revista ALAD 19(4): 146-161, 2011.
- [Background] Schinckus L, Van den Broucke S, Housiaux M; Diabetes Literacy Consortium. Assessment of implementation fidelity in diabetes self-management education programs: a systematic review. Patient Educ Couns. 2014 Jul;96(1):13-21. doi: 10.1016/j.pec.2014.04.002. Epub 2014 Apr 21. PMID 24795074
- [Background] Machado Bonfante H, da Costa Avila M, Miranda Marcon L, Andrade Pedrosa C, de Oliveira Goncalves Prince Soares H, Fonseca Reis L, Pereira Mendonca U, dos Reis Barreiros A, Porto Araújo de Andrade M. Prediabetes: Clinical Relevance of an Important Risk Marker. Revista Brasileira de Cièncias Médicas e da Saúde 3(3):1-5, 2015.
- [Background] Perez Siwik V, Kutob RM, Ritenbaugh C, Aickin M, Gordon JS. Families United/Familias Unidas: development and implementation of a family-based group office visit model for the primary prevention of type 2 diabetes. Diabetes Educ. 2012 Nov-Dec;38(6):811-21. doi: 10.1177/0145721712461533. Epub 2012 Sep 26. PMID 23019237
- [Background] Diabetes Prevention Program (DPP) Research Group. The Diabetes Prevention Program (DPP): description of lifestyle intervention. Diabetes Care. 2002 Dec;25(12):2165-71. doi: 10.2337/diacare.25.12.2165. PMID 12453955
- [Background] Lindstrom J, Louheranta A, Mannelin M, Rastas M, Salminen V, Eriksson J, Uusitupa M, Tuomilehto J; Finnish Diabetes Prevention Study Group. The Finnish Diabetes Prevention Study (DPS): Lifestyle intervention and 3-year results on diet and physical activity. Diabetes Care. 2003 Dec;26(12):3230-6. doi: 10.2337/diacare.26.12.3230. PMID 14633807
- [Background] Pan XR, Li GW, Hu YH, Wang JX, Yang WY, An ZX, Hu ZX, Lin J, Xiao JZ, Cao HB, Liu PA, Jiang XG, Jiang YY, Wang JP, Zheng H, Zhang H, Bennett PH, Howard BV. Effects of diet and exercise in preventing NIDDM in people with impaired glucose tolerance. The Da Qing IGT and Diabetes Study. Diabetes Care. 1997 Apr;20(4):537-44. doi: 10.2337/diacare.20.4.537. PMID 9096977
- [Background] Hariri S, Yoon PW, Qureshi N, Valdez R, Scheuner MT, Khoury MJ. Family history of type 2 diabetes: a population-based screening tool for prevention? Genet Med. 2006 Feb;8(2):102-8. doi: 10.1097/01.gim.0000200949.52795.df. PMID 16481893
- [Background] Kovacs Burns K, Holt RI, Nicolucci A, Lucisano G, Skovlund SE, Comaschi M, Vallis M, Peyrot M. Correlates of psychological outcomes among family members of people with diabetes in the second Diabetes Attitudes, Wishes and Needs (DAWN2() ) study. Diabet Med. 2016 Sep;33(9):1184-93. doi: 10.1111/dme.13136. Epub 2016 May 26. PMID 27086909
- [Background] Shi M, Xu MY, Liu ZL, Duan XY, Zhu YB, Shi HM, Jiang B, Zhang XM, Yu XH. Effectiveness of family involvement in newly diagnosed type 2 diabetes patients: a follow-up study. Patient Educ Couns. 2016 May;99(5):776-82. doi: 10.1016/j.pec.2015.12.018. Epub 2015 Dec 30. PMID 26763869
- [Background] Arslanian SA, Bacha F, Saad R, Gungor N. Family history of type 2 diabetes is associated with decreased insulin sensitivity and an impaired balance between insulin sensitivity and insulin secretion in white youth. Diabetes Care. 2005 Jan;28(1):115-9. doi: 10.2337/diacare.28.1.115. PMID 15616243
- [Background] Herman WH, Hoerger TJ, Brandle M, Hicks K, Sorensen S, Zhang P, Hamman RF, Ackermann RT, Engelgau MM, Ratner RE; Diabetes Prevention Program Research Group. The cost-effectiveness of lifestyle modification or metformin in preventing type 2 diabetes in adults with impaired glucose tolerance. Ann Intern Med. 2005 Mar 1;142(5):323-32. doi: 10.7326/0003-4819-142-5-200503010-00007. PMID 15738451
- [Background] Hu J, Wallace DC, McCoy TP, Amirehsani KA. A family-based diabetes intervention for Hispanic adults and their family members. Diabetes Educ. 2014 Jan-Feb;40(1):48-59. doi: 10.1177/0145721713512682. Epub 2013 Nov 18. PMID 24248832
- [Background] Mayberry LS, Harper KJ, Osborn CY. Family behaviors and type 2 diabetes: What to target and how to address in interventions for adults with low socioeconomic status. Chronic Illn. 2016 Sep;12(3):199-215. doi: 10.1177/1742395316644303. Epub 2016 Apr 19. PMID 27099387
- [Background] Kutob RM, Siwik VP, Aickin M, Ritenbaugh C. Families United/Familias Unidas: family group office visits to reduce risk factors for type 2 diabetes. Diabetes Educ. 2014 Mar-Apr;40(2):191-201. doi: 10.1177/0145721714520722. Epub 2014 Jan 24. PMID 24464087